CLINICAL TRIAL: NCT04931836
Title: The Influence of Physical Activity on the Gut Microbiome of Pre-Diabetic Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00009136
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Overweight; Overweight and Obesity; PreDiabetes; Type 2 Diabetes; Type 2 Diabetes Mellitus; Type 2 Diabetes Mellitus in Obese
Keywords: Microbiome; Physical Activity
MeSH Terms: conditions — Obesity; Overweight; Prediabetic State; Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants in this group will complete the physical activity intervention.
  Interventions: Behavioral: Physical Activity Intervention
- Control Group (No Intervention): Participants in this group will be asked to maintain their normal level of physical activity.

INTERVENTIONS:
Behavioral: Physical Activity Intervention — Three walking sessions/week for a total of 8 weeks (24 total sessions) - Walking sessions will either take place on new commercial treadmills in the Epidemiology Clinical Research Center or remotely at or around a participant's home. Regardless of the walking location, walking sessions will be 30 min in duration during intervention weeks 1 through 4 and a minimum of 45 min each during intervention weeks 5 through 8.
  Arms: Experimental Group

SUMMARY:
The present study is a 100-participant randomized controlled 2-arm parallel trial that employs a metagenomic approach to examine how 8 weeks of supervised moderate-intensity treadmill walking exercise (MWE) for 30-45 min 3 times/week alters the gut microbiome, serum short chain fatty acids, and the cardiometabolic profile, body weight, and body composition of individuals 30-64 years old who have overweight or obesity and have prediabetes.

DETAILED DESCRIPTION:
All eligible and consented participants will complete a 3-week run-in phase during which baseline outcome assessments will be performed. During run-in weeks 1 and 2, participants will wear a Fitbit Inspire 2 smartwatch and complete three unannounced dietary recalls. During the run-in week 3 (see table below), participants will consume their 3-day standardized meal plan on days three through five, obtain a fecal sample, complete a study questionnaire, and complete a study assessment visit. To quantify compliance with the 3-day meal plan, participants will be provided with a paper checklist of all foods to be consumed, and will be asked to indicate which foods were consumed and to document any deviation. The study assessment visit will include a fasting blood draw (at baseline and week eight only), blood pressure in triplicate, weight measure and body fat assessment in duplicate, and a saliva sample.

ELIGIBILITY:
Inclusion Criteria:

* Classified as overweight or obese with BMI 25.0-39.9 kg/m2.
* Documentation* of a prediabetes diagnosis within one year of enrollment by physician or primary care provider based on lab tests showing a fasted blood glucose of 100-125 mg/dL, a 2-hour oral glucose tolerance test of 140-199 mg/dL, or an HbA1c level of 5.7%-6.4%76; OR a study screening lab value of HbA1C within the afore mentioned range.
* Currently engaged in <100 min/week of physical activity - confirmed by questionnaire.
* No exercise contraindications as assessed by the Physical Activity Readiness Questionnaire (PAR-Q)78-this Questionnaire involves seven "yes" or "no" questions regarding an individual's health status, with answering "yes" to any one of these questions requiring a prospective participant to acquire a written doctor's note stating they can safely participate in the trial's exercise intervention.
* No self-reported physical/mental disabilities or gastrointestinal conditions.
* No antibiotic usage within the last 45 days.
* Stable weight over the last 6 months (<10% change).
* Not currently pregnant, planning to become pregnant, or currently breastfeeding.
* Willing to maintain current dietary and exercise habits, aside from any changes to be made per the study exercise protocol.

  * Note: Documentation can include either a print out or screen shot of the lab value illustrating eligibility, along with the date of the test and the participant's name. If a hard copy is provided, the date and name will be redacted.

Exclusion Criteria:

* Self-reported use of metformin and/or other medications that could interfere with the primary outcome.
* History of bariatric surgery or a history of other medical interventions that would interfere with the primary outcome.

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Demmer, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited on a rolling basis through a combination of the following methods: clinical referrals via partners within community-based health clinics, and fliers posted on physical (e.g. campus buildings, community billboards) and virtual (e.g. Facebook, NextDoor) walls. Finally, eligible participants based on electronic health record were identified and and invitation was sent via 'My Chart' directly to the prospective participant.
Pre-assignment Details: After consenting, participants entered a three week run-in period during which time they provided a baseline stool sample, continued regular activity, used a study provided fitbit to monitor baseline physical activity levels, and responded to three phone dietary assessments.
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 39 | 38
Completed | 35 | 37
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Three walking sessions/week for a total of 8 weeks (24 total sessions) - Walking sessions occurred remotely at or around a participant's home. Regardless of the walking location, walking sessions were 30 min in duration during intervention weeks 1 through 4 and a minimum of 45 min each during intervention weeks 5 through 8.
- Control: Participants in this group were asked to maintain their normal level of physical activity.
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 39 | 38 | 77
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.9 (9.3) | 53.1 (8.5) | 51.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 32 | 66
  Male | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 31 | 27 | 58
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 34 | 30 | 64
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: Participants]
  United States | 39 | 38 | 77
Weight (kg) [Mean (Standard Deviation); unit: Kilogram] — Weight in Kg
  Kilogram | 99 (21.5) | 97.1 (19.6) | 98.1 (20.5)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 34.7 (6.1) | 34.1 (5.4) | 34.4 (5.7)
Percent body fat [Mean (Standard Deviation); unit: %] | 44.0 (7.2) | 43.5 (6.7) | 43.8 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Shannon Index (Unitless)
Description: Changes to the gut microbiome will be assessed via metagenomic sequencing, from pre- to post-intervention. The Shannon Index-a measure of microbial community diversity-will be the primary indicator for changes in gut microbiota composition, and will be assessed at baseline, and following the 4th and 8th weeks. Index values are unitless and range from 0 to 1. Lower values indicate more diversity while higher values indicate less diversity. Outcome will be reported at baseline, 4 weeks, and 8 weeks and as the change from baseline to 4 weeks and baseline to 8 weeks.
Time Frame: 8 weeks
Population: There were 6 participants with missing microbiome data.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 35 | 36
units on a scale | -0.20 (.073) | 0.013 (.072)

2. Primary Outcome: Change in Serum Short Chain Fatty Acids (SCFA)
Description: Participants will undergo fasted blood draws to assess serum SCFA levels. This work will be performed using the Metabolon pipeline. Outcome is reported as the sum of the serum concentrations of acetate, propionate, and butyrate in Z-score units. We report the Week 8 means and standard errors from a linear model adjusted for the Week 0 (baseline) values. The original units are reported in ng/mL and the final results are reported as standardized z-scores in which each value subtracts the mean and the difference is divided by the standard deviation. Higher values represent higher levels of SCFA which is considered better. The scale is in standard deviation units. A value of 0 = the population mean.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 33 | 37
score on a scale | 0.19 (0.107) | 0.08 (0.101)

3. Secondary Outcome: High-density Lipoprotein Cholesterol (HDL-C)
Description: High-density lipoprotein cholesterol (HDL-C) will be measured using standard laboratory test and report in units of mg/dl. We report the Week 8 means and standard errors from a linear model adjusted for the Week 0 (baseline) values.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Intervention | Control
Number analyzed (Participants) | 33 | 37
mg/dL | 53.4 (0.73) | 51.7 (0.69)

4. Secondary Outcome: Triglycerides
Description: Blood triglycerides will be measured using a standard laboratory test and reported in units of mg/dl. We report the Week 8 means and standard errors from a linear model adjusted for the Week 0 (baseline) values.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Intervention | Control
Number analyzed (Participants) | 33 | 37
mg/dL | 147.2 (7.08) | 142.7 (6.70)

5. Secondary Outcome: Fasting Insulin
Description: Fasting insulin will be measured by laboratory test and reported in units of pm/ml. We report the Week 8 means and standard errors from a linear model adjusted for the Week 0 (baseline) values.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: pm/L
Arm/Group | Intervention | Control
Number analyzed (Participants) | 32 | 36
pm/L | 132.5 (8.96) | 134.8 (8.44)

6. Secondary Outcome: Fasting Glucose
Description: Fasting glucose will be measured by standard laboratory test and reported in units of mg/dl. We report the Week 8 means and standard errors from a linear model adjusted for the Week 0 (baseline) values.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Intervention | Control
Number analyzed (Participants) | 33 | 36
mg/dL | 105.0 (1.42) | 105.0 (1.35)

7. Secondary Outcome: C-reactive Protein (CRP)
Description: C-reactive protein (CRP) will be measured by laboratory test and reported in units of mg/l. We report the Week 8 means and standard errors from a linear model adjusted for the Week 0 (baseline) values.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Intervention | Control
Number analyzed (Participants) | 31 | 37
mg/L | 4.6 (0.36) | 4.5 (0.33)

8. Secondary Outcome: Resting Systolic Blood Pressure (BP)
Description: Resting systolic blood pressure will be reported in units of mmHg. We report the Week 8 means and standard errors from a linear model adjusted for the Week 0 (baseline) values.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Intervention | Control
Number analyzed (Participants) | 34 | 36
mmHg | 121 (1.9) | 120 (1.8)

9. Secondary Outcome: Body Composition
Description: Body composition will be analyzed using bioelectrical impedance. Outcome will be reported as percent body fat. We report the Week 8 means and standard errors from a linear model adjusted for the Week 0 (baseline) values.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 34 | 36
Percentage | 43.5 (0.41) | 43.6 (0.40)

10. Secondary Outcome: Cardiometabolic Risk Score (CMR)
Description: The Cardiometabolic Risk Score (CMR) is the mean Z-score across systolic blood pressure, glucose, insulin, HDL, % body fat, and triglycerides. We report the Week 8 means and standard errors from a linear model adjusted for the Week 0 (baseline) values. The final results are reported as standardized z-scores in which each value subtracts the mean and the difference is divided by the standard deviation. Higher values represent higher levels of cardiometabolic risk which is considered worse. The scale is in standard deviation units. A value of 0 = the population mean.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: z-score standardized units
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 30 | 35
z-score standardized units | -.01 (.050) | -.04 (.047)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/38
Other Adverse Events (participants affected / at risk) | 0/39 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/36/NCT04931836/Prot_SAP_000.pdf